CLINICAL TRIAL: NCT05650255
Title: A Digital Twin for Exoskeleton Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202209051RINB
Record Dates: First submitted 2022-11-27; First posted 2022-12-14 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Human Intention; Exoskeletons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Digital Twin for Exoskeleton Pilot (Experimental): This project is expected to use different machine learning models to make accurate predictions of human intent when healthy people drive different actions or action transitions of common human actions. Drivers will wear sensors such as inertial measurement unit (IMU) and electromyography (EMG) in the lower limbs to measure body signals of participants during actions in a non-invasive way, and let the system calculate the joint angle, angular velocity and angular acceleration of each joint of the driving lower limb related human signals.
  Interventions: Other: A Digital Twin for Exoskeleton Pilot

INTERVENTIONS:
Other: A Digital Twin for Exoskeleton Pilot — The purpose of this project is to establish a digital twin of this driving, which will perform the driving action in parallel, and calculate in parallel in the virtual environment the torque required to provide each joint torque to maintain stable walking without falling, and this torque can be used as a monitoring basis for the auxiliary torque of each axis for the exoskeleton. When the exoskeleton's movements are out of range of a stable gait, the controller can warn and attenuate the output of auxiliary forces, and on the other hand, it has the opportunity to analyze whether the intention of driving is to switch the movement mode - such as stopping, or sitting, squatting, etc.

SUMMARY:
Although exoskeletons have been studied for many years, actual products have been sold on the market. However, there are still many limitations in the practical application of exoskeletons, and the control logic is also limited to the level of motor torque compensation, and lacks the consideration of overall motion stability (such as whether the wearer (driving, pilot) will fall). The purpose of this project is to establish a digital twin of this driving, which will perform the driving action in parallel, and calculate in parallel in the virtual environment the torque required to provide each joint torque to maintain stable walking without falling, and this torque can be used as a monitoring basis for the auxiliary torque of each axis for the exoskeleton. When the exoskeleton's movements are out of range of a stable gait, the controller can warn and attenuate the output of auxiliary forces, and on the other hand, it has the opportunity to analyze whether the intention of driving is to switch the movement mode - such as stopping, or sitting, squatting, etc.

DETAILED DESCRIPTION:
This project is expected to use different machine learning models to make accurate predictions of human intent when healthy people drive different actions or action transitions of common human actions. Drivers will wear sensors such as inertial measurement unit (IMU) and electromyography (EMG) in the lower limbs to measure body signals of participants during actions in a non-invasive way, and let the system calculate the joint angle, angular velocity and angular acceleration of each joint of the driving lower limb related human signals.

ELIGIBILITY:
Inclusion Criteria:

1. Can stand independently and walk for more than 5 minutes.
2. According to age, it can be divided into: elderly groups (aged between 50~80 years old); Young people (aged 18~50 years).

Exclusion Criteria:

1. Have current or previous neurological diseases of the lower extremities, such as: acute neuritis, stroke, Parkinson's disease.
2. Have current or previous orthopedic diseases of the lower extremities, such as: knee replacement, rheumatoid arthritis, or sports injuries and other symptoms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The angles of the subject's joints. | 3 years
  The angles of the subject's joints (unit: degree) are performed by using IMU sensors when subjects do some action such as standing, walking or sitting.
The activities of muscles state of human movement. | 3 years
  The activities of muscles state of human movement (unit: millivolt or %) are performed by using EMG sensors when subjects do some action such as standing, walking, sitting, squatting or step-up.
The comprehensive intention of the subjects. | 3 years
  The comprehensive intention time of the human body (unit: second) is performed by using IMU sensors and EMG sensors when subjects do some action such as standing, walking, sitting, squatting or step-up.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Hsu, Ph.D, Study Director — Study Principal Investigator National Taiwan Unversity
Locations (1):
- National Taiwan University Hospital, Taipei,Taiwan, Taiwan